CLINICAL TRIAL: NCT05130606
Title: Testing a Narrative Intervention to Enhance Genetic Counseling and Testing
Brief Title: CONTIGO - A Narrative Intervention to Enhance Genetic Counseling and Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002789; 1R01CA248543-01A1 (NIH)
Record Dates: First submitted 2021-09-07; First posted 2021-11-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Breast and Ovarian Cancer
Keywords: Breast cancer; Ovarian cancer; Hereditary cancer; Latinas
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Hybrid Type 1 research design (efficacy study). Two arm randomized controlled trial and Implementation Focused Process Evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Arm (Experimental): Culturally Targeted Narrative Video: "Is My Cancer Hereditary? Rosa Visits a Genetic Counselor." Participants in the video arm will be asked to watch an 18-minute video that the research team developed and tested previously about HBOC and genetic services. The video is recorded with Spanish audio and is available with English subtitles.
  Interventions: Behavioral: Culturally Targeted Narrative Video: "Is My Cancer Hereditary? Rosa Visits a Genetic Counselor."
- Fact Sheet Arm (Active Comparator): Participants in the Fact Sheet arm will receive a Fact sheet about HBOC and genetic services and will be asked to read it in their own time. The Fact Sheet is available in English and Spanish.
  Interventions: Behavioral: FORCE Fact Sheet

INTERVENTIONS:
Behavioral: Culturally Targeted Narrative Video: "Is My Cancer Hereditary? Rosa Visits a Genetic Counselor." — Participants randomized to the video arm will receive a link with a password by email or text message to watch the video, depending on participants' preference. Participants without internet access will receive a DVD. Participants will be instructed to watch the video alone with no interruptions. We will ask them not to share the link with others.
  Arms: Video Arm
Behavioral: FORCE Fact Sheet — Participants will receive a PDF of the fact sheet by email, text message, or a printed fact sheet by mail depending on participants' preferences. The fact sheet includes information about genes, breast cancer, risk factors for HBOC, genetic counseling and testing, and resources.
  Arms: Fact Sheet Arm

SUMMARY:
This is a mixed-methods Hybrid Type 1 research design (efficacy study) in which we aim to conduct a two-arm randomized controlled trial and an Implementation Focused Process Evaluation of a culturally-targeted video and referral screening tool.

In this study, the investigators aim to evaluate the efficacy of a culturally targeted video previously developed by the research team vs. a Spanish-language fact sheet from an established group on enhancing genetic counseling and testing uptake and psychosocial outcomes in Latina women at risk for hereditary breast and ovarian cancer.

The investigators will test the video's efficacy while also gathering data on the implementation and future sustainability of using the Risk Screening Tool (RST) and video in community clinics.

DETAILED DESCRIPTION:
The investigators previously developed and piloted a culturally targeted narrative video in Spanish to provide HBOC and GCT education to at-risk Latinas. The investigators expanded traditional approaches to address psychosocial barriers through risk messages designed to elicit emotional responses; emotions are often stronger predictors of behavior than cognition. Our video is responsive to Latinas' preferences, targets motivators, and addresses psychosocial barriers identified in our formative research.

In this study, the investigators aim to evaluate the efficacy of our video vs. a fact sheet from an established group on enhancing GCT uptake and psychosocial outcomes on a two-arm randomized controlled trial. The investigators will test the video's efficacy while also gathering data on the implementation and future sustainability of using an adapted Risk Screening Tool (RST) and video in community clinics.

The investigators will partner with community clinics and implement a Risk Screening Tool (RST) at their practice to identify women at risk of HBOC. Community clinic staff (N~32) will be asked to participate in a pre-implementation and a post-implementation focus group to assess implementation outcomes of integrating HBOC screening practices in their clinic. Through the community clinics, the investigators aim to recruit N~300 Latina women at risk for HBOC based on their personal or family history of cancer. Latina women at risk for HBOC will be randomized to a Video arm or Fact Sheet Arm. All participants in the randomized controlled trial will be offered genetic counseling and testing.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 and 2.

* Self-identify as a Latina woman
* Be 18 years old or older
* Be able to provide informed consent
* Be fluent in Spanish
* Meet NCCN criteria to be considered for genetic cancer risk assessment for HBOC, whether by a personal history of cancer or family history of cancer
* No previous participation in genetic counseling or testing for hereditary breast and ovarian cancer risk
* No other family members are participating in this study
* Have not participated in any previous studies involving interventions about HBOC or GCT

Aim 3.

* Be 18 years old or older
* Be fluent in English or Spanish
* Have a role in the partner community clinic as either a) full-time or part-time employee b) intern c) volunteer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only self-identified women will be recruited for this study
Enrollment: 332 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of Genetic Counseling | Change from the baseline survey to four months after baseline
  Participants will self report whether they attended a genetic counseling session in the four months following their baseline survey. The study team will also have direct access to the genetic counseling company's records.
Uptake of Genetic Testing | Change from the baseline survey to four months after baseline
  Participants will self report whether they completed a genetic test for hereditary cancer in the four months following their baseline survey. The study team will also have direct access to the genetic counseling company's records.

SECONDARY OUTCOMES:
Knowledge about HBOC | Change from the baseline to two-week after baseline, and change from two-week follow up survey to four months after baseline
  9-item Scale from Kasting et al, 2019. The scale has statements to which participants respond True, False, or I don't Know. The scale is scored based on the accuracy of responses. A higher score indicates higher knowledge. Scores range from 0-9.
Self-efficacy about attending genetic cancer risk assessment | Change from the baseline to two-week after baseline
  Change in self-efficacy about genetic counseling and testing will be measured by specific items from the Theory of Planned Behavior scale (Ajzen, 2002) on a scale from 1-7 -Not at all to 7- Extremely)
Beliefs and Attitudes about genetic cancer risk assessment | Change from the baseline to two-week after baseline
  Changes in beliefs and attitudes about genetic counseling and genetic testing. The outcome will be assessed by 22 items from a scale developed by Sussner, Jandorf, Thompson et al., 2012 in which participants respond to a Likert-type scale from 1 (completely disagree) to 7 (completely agree).
Subjective norms about genetic cancer risk assessment | Change from the baseline to two-week after baseline
  Change in subjective norms about genetic counseling and testing will be measured by specific items from the Theory of Planned Behavior scale (Ajzen, 2002) on a scale from 1-Not at all to 7- Extremely)
Anticipatory emotions about genetic cancer risk assessment | Change from the baseline to two-week after baseline
  Scale items on a 7-point Likert-type response (from 1-strongly disagree to 7-strongly agree).
Acceptability of the intervention | At two weeks after baseline
  Overall acceptability is measured on a 4-item self-reported scale ranging from 1 to 10, where 1 = not at all to 10 = highly
Feasibility of the intervention | At two weeks after baseline
  Proportion of women who have watched/read the video or fact sheet at the two week follow up

OTHER OUTCOMES:
Feasibility of the Referral Screening Tool | Change from the pre-implementation focus groups with community clinics to post implementation focus groups with community clinics (48 months)
  Qualitative measure captured through semi-structured interviews using the Consolidated Framework for Implementation Research. (e.g., What barriers and facilitators did you experience while implementing the RST?)
Acceptability of the Referral Screening Tool | Change from the pre-implementation focus groups with community clinics to post implementation focus groups with community clinics (48 months)
  Qualitative measure captured through semi-structured interviews using the Consolidated Framework for Implementation Research.
Adoption of the Referral Screening Tool | At the post implementation focus groups with community clinics adoption over the previous 48 months will be assessed
  Qualitative measure captured through semi-structured interviews using the Consolidated Framework for Implementation Research.
Sustainability of the Referral Screening Tool | At the post implementation focus groups with community clinics sustainability of the screener based on their experience during the previous 48 months will be assessed
  Qualitative measure captured through semi-structured interviews using the Consolidated Framework for Implementation Research.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Hurtado de Mendoza, Ph.D, Principal Investigator — Georgetown Lombardi Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No